CLINICAL TRIAL: NCT04293614
Title: Invasive Arterio-Venous Fistula Blood Pressure Monitoring & Fluid Dynamics Study
Status: Completed | Type: Observational
Sponsor: University Hospital of Limerick (Other)
Collaborators: University of Limerick (Other)
Responsible Party: Principal Investigator, Fiona Leahy, Professor Eamon Kavanagh Prinicipal Investigator, University Hospital of Limerick
Other Study IDs: DVS005
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Arterio-venous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The surgical formation of an AVF offers a unique example of vascular remodelling and adaption. Yet, the specific factors which elicit remodelling events which determine successful maturation or failure have not been unambiguously determined.

Computational fluid dynamic (CFD) simulations are increasingly been employed to investigate the interaction between local haemodynamics and remodelling and can potentially be used to assist in clinical risk assessment of maturation or failure.

However, these simulations are inextricably linked to their prescribed boundary conditions and are reliant on in vivo measurements of flow and pressure to ensure their validity. This study will compare in vivo measurements of the pressure distribution across an AVF against a representative numerical model.

DETAILED DESCRIPTION:
Most patients with End Stage Renal Disease (ESRD) will require haemodialysis. Several studies have recognized a well-functioning Arterio-Venous Fistula (AVF) as the best modality for access in patients with ESRD undergoing haemodialysis.

A mature AVF has lower incidence of thrombosis and stenosis compared to the other two available modalities of the Arterio-Venous Graft (AVG) and Central Venous Catheter (CVC). This translates into prolonged patency rates and lower risk of infection. The use of AVF's are also associated with lower mortality, and costs.

However, significant numbers of AVFs [20% to 60 %] are known to fail to mature into functioning fistulas. Issues such as impaired vein remodelling, intimal hyperplasia, technical problems, unrecognized stenosis within the outflow vein, inflow problems, or steal syndromes can all lead to failure of achieving a mature AVF.

The aim of the study is to examine the relationship between the pressure gradient within the surgically formed AVF and its' maturation and functioning status.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing AVF formation surgical procedure or AVF intervention surgery.
2. Willing and capable of signing an informed consent form.

Exclusion Criteria:

1. Patients unable to provide informed consent.
2. Patients under the age of 18
3. Patients who are deemed unsuitable due to any circumstances as deemed appropriate by the P.I.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of individuals with ESRD who are undergoing AVF creation or intervention surgery for the purpose of undergoing Haemodialysis treatment.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-01-14 (Actual)

PRIMARY OUTCOMES:
Effects of pressure gradient within AVF on maturation and functioning of the AVF. | 2 years
  Pressure measurements obtained intra-operatively will be examined alongside pre and post operative ultrasound imaging of the veins and arteries.

SECONDARY OUTCOMES:
Comparison of in-vivo and ex-vivo perfusion with validation of CFD solutions. | 2 years
  The two models will be compared for validation purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Eamon Kavanagh, MD FRCSI, Principal Investigator — University Hospital of Limerick
Locations (1):
- University Hospital Limerick, Limerick, Ireland

IPD SHARING:
Plan to Share IPD: Undecided